CLINICAL TRIAL: NCT02483702
Title: The Affect of Radiated Versus Non-Irradiated Blood on Extracellular Potassium Levels in Infants Undergoing Craniosynostosis Repair
Brief Title: Irradiated Blood Versus Non Irradiated Blood Transfusions in Craniosynostosis Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valley Anesthesiology Consultants (Other)
Responsible Party: Principal Investigator, Neil Raj Singhal, Director of Research, Valley Anesthesiology Consultants
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15-063
Record Dates: First submitted 2015-06-22; First posted 2015-06-29 (Estimated); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Graft Versus Host Disease; Hyperkalemia; Craniectomy; Synostectomy; FOA; Congenital Malformations
Keywords: Irradiated Blood; Non-Irradiated Blood; graft versus host disease; TA-GVHD; potassium; Blood transfusion
MeSH Terms: conditions — Graft vs Host Disease; Hyperkalemia; Congenital Abnormalities

ARMS (2):
- Patients under 4 months Receive Irradiated Blood (Experimental): Patients under 4 months of age will receive irradiated blood products, as per hospital protocol. The patient's extracellular potassium levels will be recorded pre-transfusion, at 30 minute intervals during the transfusion, and post-transfusion. The collected data will be compared to test for correlation between extracellular potassium levels, the type of blood transfused, and the amount of calcium that is administered.
  Interventions: Other: Irradiated Blood Transfusions
- Patients Over 4 Months Recieve Non-Irradiated Blood (Experimental): Patients over 4 months of age will receive non-irradiated blood products. The patient's extracellular potassium levels will be recorded pre-transfusion, at 30 minute intervals during the transfusion, and post-transfusion. The collected data will be compared to test for correlation between extracellular potassium levels, the type of blood transfused, and the amount of calcium that is administered.
  Interventions: Other: Non-Irradiated Blood Transfusions

INTERVENTIONS:
Other: Irradiated Blood Transfusions — Same as arm description - need to collect extracellular potassium values.
  Arms: Patients under 4 months Receive Irradiated Blood
Other: Non-Irradiated Blood Transfusions — Same as arm description - need to collect extracellular potassium values.
  Arms: Patients Over 4 Months Recieve Non-Irradiated Blood

SUMMARY:
Blood transfusions are required for patients undergoing a craniosynostosis repair due to the significant amount of blood loss. Irradiated or non-irradiated transfusions have many risks involved including elevated potassium levels and graft versus host disease (TA-GVHD). Irradiated blood is able to destroy the leukocytes responsible for TA-GVHD, but it adversely causes elevated extracellular potassium due to hemolysis of the RBC's. When this blood is transfused, it may introduce too much extracellular potassium (> 6.5 meq/L) into the patient causing interference with the heart's conduction system significantly increasing the risk for hemodynamic changes, cardiac arrhythmias, and cardiac arrest. Hyperkalemia from rapid transfusions occurs much more frequently than TA-GVHD; however, both complications are under-reported.

The study aims to evaluate the risk of irradiated versus non-irradiated blood in patients under the age of 6 months undergoing a craniosynostosis repair. This will be done by comparing the levels of extracellular potassium pre-transfusion, during transfusion, immediately after transfusion, and 30 minutes after the completion of transfusion. The investigators hypothesize that the patients who receive irradiated blood will have an increased extracellular potassium level compared to those who receive non-irradiated blood.

DETAILED DESCRIPTION:
Patients between the ages of 2 to 6 months of age and undergo a sagittal synostosis repair will split into two groups to participate in a prospective pilot study. The purpose of this study is to examine the extracellular potassium levels in patients who receive irradiated blood versus non-irradiated blood. Enrollment will occur over a 24 month period or until 20 patients are enrolled. The patient names, medical record numbers and any other identifiers will be kept strictly confidential.

Patients will receive irradiated or non-irradiated blood based on their age. Patients under 4 months of age will receive irradiated blood products, as per hospital protocol, while patients over 4 months of age will receive non-irradiated blood products.

Patients will receive standard surgical practice for their craniosynostosis repair and will receive the blood transfusion at the discretion of the anesthesiologist and surgeon. All the blood that is transfused will be analyzed prior to transfusion. The patient's extracellular potassium levels will be recorded pre-transfusion, at 30 minute intervals during the transfusion, and post-transfusion. The collected data will be compared to test for correlation between extracellular potassium levels, the type of blood transfused, and the amount of calcium that is administered.

There is minimal risk of harm associated with the study. All surgical procedures run their typical risk of infection, bleeding or any other complication that could occur during or after the operation. The blood transfusions may also increase patient's risk of graft versus host disease, hyperkalemia, or cardiac anomalies. These cases will be documented and responded to according to anesthesiologist and surgeon's preference.

Materials and information necessary to carry out this experiment include: patient age, sex, weight, type of blood transfused (ABO and non-irradiated/irradiated), vital signs, operating time, amount of blood lost, adverse events, and length of stay.

Patients who decline participation in the study will have no change in their anesthetic or post-operative care.

ELIGIBILITY:
Inclusion Criteria:

* Must be between 2-6 m/o
* Must be undergoing a craniosynostosis repair
* Must require a blood transfusion

Exclusion Criteria:

* n/a

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2015-08; Primary Completion 2017-05-11 (Actual); Study Completion 2017-05-11 (Actual)

PRIMARY OUTCOMES:
Change in extracellular potassium values. | immediately after transfusion and 30 minutes after the end of transfusion
  We hope to determine if irradiated blood will pose a greater risk for hyperkalemia than non-irradiated blood products. This will be done by looking at potassium values immediately after transfusion and again 30 minutes after the end of transfusion.

CONTACTS AND LOCATIONS:
Locations (1):
- Phoenix Children's Hospital, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharma S, Sharma P, Tyler LN. Transfusion of blood and blood products: indications and complications. Am Fam Physician. 2011 Mar 15;83(6):719-24. PMID 21404983
- [Background] Rosen NR, Weidner JG, Boldt HD, Rosen DS. Prevention of transfusion-associated graft-versus-host disease: selection of an adequate dose of gamma radiation. Transfusion. 1993 Feb;33(2):125-7. doi: 10.1046/j.1537-2995.1993.33293158043.x. PMID 8430450
- [Background] Schroeder ML. Transfusion-associated graft-versus-host disease. Br J Haematol. 2002 May;117(2):275-87. doi: 10.1046/j.1365-2141.2002.03450.x. No abstract available. PMID 11972509
- [Background] Lee AC, Reduque LL, Luban NL, Ness PM, Anton B, Heitmiller ES. Transfusion-associated hyperkalemic cardiac arrest in pediatric patients receiving massive transfusion. Transfusion. 2014 Jan;54(1):244-54. doi: 10.1111/trf.12192. Epub 2013 Apr 15. PMID 23581425
- [Background] Bontadini A, Tazzari PL, Manfroi S, Tassi C, Conte R. Apoptosis in leucodepleted packed red blood cells. Vox Sang. 2002 Jul;83(1):35-41. doi: 10.1046/j.1423-0410.2002.00191.x. PMID 12100387
- [Background] Weiskopf RB, Schnapp S, Rouine-Rapp K, Bostrom A, Toy P. Extracellular potassium concentrations in red blood cell suspensions after irradiation and washing. Transfusion. 2005 Aug;45(8):1295-301. doi: 10.1111/j.1537-2995.2005.00220.x. PMID 16078915
- [Background] Olson J, Talekar M, Sachdev M, Castellani W, De la Cruz N, Davis J, Liao J, George M. Potassium changes associated with blood transfusion in pediatric patients. Am J Clin Pathol. 2013 Jun;139(6):800-5. doi: 10.1309/AJCP2MP8OIIXNKXF. PMID 23690124
- [Background] Vraets A, Lin Y, Callum JL. Transfusion-associated hyperkalemia. Transfus Med Rev. 2011 Jul;25(3):184-96. doi: 10.1016/j.tmrv.2011.01.006. Epub 2011 Apr 17. PMID 21498041
- [Background] Faberowski LW, Black S, Mickle JP. Blood loss and transfusion practice in the perioperative management of craniosynostosis repair. J Neurosurg Anesthesiol. 1999 Jul;11(3):167-72. doi: 10.1097/00008506-199907000-00002. PMID 10414670